CLINICAL TRIAL: NCT04452734
Title: Efficacy of Platelet Rich Plasma (PRP) on Mouth Opening and Pain After Surgical Extraction of Mandibular Third Molars.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2020/3
Record Dates: First submitted 2020-04-06; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-04

CONDITIONS: Tooth Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Procedure: Surgical Extraction
- Study Group (Experimental)
  Interventions: Procedure: Platelet Rich Plasma (PRP); Procedure: Surgical Extraction

INTERVENTIONS:
Procedure: Platelet Rich Plasma (PRP) — PRP was prepared by withdrawing 8-10 ml of patients own blood (IV from antecubiodal area and collected in a vacuum tube coated with anticoagulant (Na citrate). For activation 1 ml of calcium chloride was added to Platelet Rich Plasma. This layer of approximately 2 ml of PRP was then taken into the residual bone cavity along with gel sponge to stimulate regeneration in wound healing after surgical extraction of mandibular third molar tooth followed by sutures
  Arms: Study Group
Procedure: Surgical Extraction — Surgical extraction procedure under Local anesthesia on dental chair, followed by spongstone (gel sponge) and suture placement.

SUMMARY:
Wisdom tooth extraction is the most common surgical procedure being carried out in oral surgical departments. The complications carried by post operative period include pain and trismus and may affect patient's quality of life.

PRP is an autologous concentrate of platelet in plasma and accelerate healing by production of growth factors. PRP is prepared from patient's own blood and later packed with gel sponge (Spongistone) in the experimental group immediately after surgical extraction of mandibular third molar teeth, followed by suture placement to close the surgical site.

DETAILED DESCRIPTION:
Wisdom tooth extraction is the most common surgical procedure being carried out in oral surgical departments. The complications carried by post operative period includes pain, swelling, trismus , along with disturbance in post extraction wound healing which may significantly affect patient's quality of life.

PRP is an autologous concentrate of platelet suspended in plasma and accelerate healing by production of various growth factors. PRP is prepared from patient's own blood and later packed with gel sponge (Spongistone) in the experimental group immediately after surgical extraction of mandibular third molar teeth, followed by suture placement to close the surgical site. PRP speeds up healing by concentration of growth factors which can lessen the inflammation and decreases trismus and pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-45 iyears
2. Either gender
3. Patients requiring extraction of mandibular 3rd molars
4. ASA grade1
5. Nonsmokers & non alcoholics
6. Not allergic to any medicines
7. No pain before the extraction procedure
8. No trismus, i.e. normal mouth opening before the extraction procedure -

Exclusion Criteria:

a) Systemic diseases b) Compromised immune system c) Platelet count less than 1.5 lacs/cmm d) Allergy to drugs e) Patients not willing to participate in the study f) Pregnant females/Lactating mothers g) Presence of pericoronitis, periapical infection or any associated lesion.

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2016-05-14 (Actual); Study Completion 2016-05-14 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 1 day
  Visual Analogue Scale (VAS) used to quantify pain
Visual Analogue Scale (VAS) | 3rd post op day
  Visual Analogue Scale (VAS) used to quantify pain
Visual Analogue Scale (VAS) | 7th post op day
  Visual Analogue Scale (VAS) used to quantify pain
Trismus | 1 day
  Trismus was quantified/measured using Vernier Calliper.
Trismus | 3rd post op day
  Trismus was quantified/measured using Vernier Calliper.
Trismus | 7th post op day
  Trismus was quantified/measured using Vernier Calliper.

CONTACTS AND LOCATIONS:
Overall Officials: Maidah Hanif, BDS, FCPS, Principal Investigator — Foundation University College of Dentistry; Muhammad Azhar Sheikh, BDS, MSc, FFD, Study Chair — Foundation University College of Dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogundipe OK, Ugboko VI, Owotade FJ. Can autologous platelet-rich plasma gel enhance healing after surgical extraction of mandibular third molars? J Oral Maxillofac Surg. 2011 Sep;69(9):2305-10. doi: 10.1016/j.joms.2011.02.014. Epub 2011 May 7. PMID 21550158
- [Background] Celio-Mariano R, de Melo WM, Carneiro-Avelino C. Comparative radiographic evaluation of alveolar bone healing associated with autologous platelet-rich plasma after impacted mandibular third molar surgery. J Oral Maxillofac Surg. 2012 Jan;70(1):19-24. doi: 10.1016/j.joms.2011.03.028. Epub 2011 Jul 20. PMID 21778014